CLINICAL TRIAL: NCT07162883
Title: A Randomized, Double-Blind, Multicenter, Pharmacokinetic Equivalence Clinical Trial of QL2107 (Keytruda® Biosimilar Candidate) in Comparison With Keytruda® (Pembrolizumab) for Adjuvant Therapy to Demonstrate Pharmacokinetic Similarity in Subjects With Resected Non-Small Cell Lung Cancer
Brief Title: Pharmacokinetic Study of QL2107 Versus Keytruda® for Adjuvant Therapy of Non-Small Cell Lung Cancer (NSCLC)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL2107-102; 2024-519883-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Neoplasm Metastasis; Neoplastic Processes; Pathologic Processes; Lung Neoplasms; Lymphatic Metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Neoplasm Metastasis; Neoplastic Processes; Pathologic Processes; Lung Neoplasms; Lymphatic Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL2107 200mg (Experimental): Participants will receive QL2107 200 milligrams (mg) intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21 days treatment cycle for up to 17 treatment cycles.
  Interventions: Drug: QL2107
- Keytruda® 200 mg (Active Comparator): Participants will receive Keytruda® 200 mg IV infusion Q3W, on Day 1 of each 21- days treatment cycle for up to 17 treatment cycles.
  Interventions: Drug: Keytruda®

INTERVENTIONS:
Drug: QL2107 — IV infusion.
  Arms: QL2107 200mg
Drug: Keytruda® — IV infusion.
  Arms: Keytruda® 200 mg

SUMMARY:
The primary purpose of this study is to demonstrate Pharmacokinetic similarity in exposure after the initial dose and at steady state of QL2107 compared with Keytruda.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (male or female) more than and equal to 18 years of age on the day of signing the ICF.
* Disease status: Participants with completely resected, histologically- or cytologically-confirmed (Stage II or IIIA) NSCLC
* Treatment with platinum-based chemotherapy; • Chemotherapy must have begun within 12 weeks after the resection surgery. The last chemotherapy dose must have been completed at least 3 weeks and no more than 12 weeks before the participant is randomized.
* No evidence of disease (NSCLC) for the post-surgery baseline assessment must be documented by full chest/abdomen/pelvis computed tomography (CT) and/or magnetic resonance imaging (MRI) and brain CT/MRI within 12 weeks prior to the randomization date.
* Eastern Cooperative Oncology Group performance status of 0 or 1.

Exclusion Criteria:

* Surgical-related adverse events (AEs) or chemotherapy-related toxicity not resolved to Grade 1, with the exception of Grade <=2 alopecia, fatigue, neuropathy, and lack of appetite/nausea.
* Participants who have received systemic corticosteroids (more than [>] 10 mg prednisone daily or equivalent) or other immunosuppressive drugs (such as cyclophosphamide, azathioprine, methotrexate, thalidomide, or tumor necrosis factor alpha inhibitors) within 2 weeks prior to the first dose.
* Participants with known epidermal growth factor receptor (EGFR)-sensitive mutations or anaplastic lymphoma kinase (ALK) gene translocations are not allowed.
* Received prior therapy with an anticytotoxic T-lymphocyte antigen-4 mAb (example, ipilimumab); anti-programmed cell death 1 (PD-1), anti-programmed cell death ligand 1 (Programmed Death-Ligand 1), or anti-programmed cell death ligand 2 (PD-L2) agent; or agent directed to another stimulatory or co-inhibitory T cell receptor.
* Participants with any active autoimmune disease or history of autoimmune diseases including but not limited to autoimmune hepatitis, interstitial pneumonia, pulmonary fibrosis, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
AUCtau,sd of QL2107 and Keytruda | At Cycle 1 (cycle length = 21 days)]
  Area under the concentration time curve for 1 dosing interval (tau = 21 days) after a single initial) dose (AUCtau,sd) of QL2107 and Keytruda® will be reported.
AUCtau,ss of QL2107 and Keytruda | At Cycle 7 (cycle length = 21 days)]
  Area under the concentration time curve for 1 dosing interval (tau = 21 days) at steady state (AUCtau,ss) of QL2107 and Keytruda® will be reported.

SECONDARY OUTCOMES:
Cmax,sd of QL2107 and Keytruda | At Cycle 1 (cycle length = 21 days)]
  Maximum (peak) serum concentration after a single dose (Cmax,sd) of QL2107 and Keytruda® will be reported.
Cmax,ss of QL2107 and Keytruda | At Cycle 7 (cycle length = 21 days)]
  Maximum (peak) serum concentration at steady state (Cmax,ss) of QL2107 and Keytruda® will be reported.
Ctrough of QL2107 and Keytruda | Up to Cycle 10 at Predose (cycle length = 21 days)
  The trough serum concentration measured before the next dose is administered (Ctrough) of QL2107 and Keytruda® (predose samples) will be reported.
Number of Participants With Antidrug Antibodies (ADAs) and Neutralizing Antibodies (NAbs) | Up to Week 52
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to Week 52

IPD SHARING:
Plan to Share IPD: No